CLINICAL TRIAL: NCT06210113
Title: The Effectiveness of Mindfulness-based Stress Reduction (MBSR) Programme for Parents of Children With ADHD: a Pilot Randomized Controlled Trial
Brief Title: Training Parents of Children With ADHD by Mindfulness-based Stress Reduction for Reducing Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: The Salvation Army, Hong Kong and Macau Command (Other)
Responsible Party: Principal Investigator, Yim Wah MAK, Ph.D, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HSEARS S20211015010
Record Dates: First submitted 2023-12-20; First posted 2024-01-18 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Stress, Psychological
Keywords: Mindfulness-based stress reduction, parental stress, Attention-Deficit Hyperactivity Disorder ADHD; parent
MeSH Terms: conditions — Stress, Psychological; Attention Deficit Disorder with Hyperactivity | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Intervention Model Description: MBSR intervention
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness (Experimental): 8-week mindfulness-based stress reduction training
  Interventions: Behavioral: Mindfulness-based Stress Reduction
- Placebo (No Intervention): received usual care

INTERVENTIONS:
Behavioral: Mindfulness-based Stress Reduction — An 8-week Mindfulness-based stress reduction training programme
  Arms: Mindfulness

SUMMARY:
The study aimed at comparing the effects of 8-week MBSR programme intervention group with usual care group in reducing parental stress and improving quality of life of parents of children with ADHD in Chinese culture.

DETAILED DESCRIPTION:
This study aimed at comparing the effects of 8-week mindfulness-based stress reduction (MBSR) intervention with usual care in improving the parental stress, quality of life, and the feasibility and acceptability of MBSR of parents of children with Attention Deficit Hyperactivity Disorder (ADHD) in Chinese context after the coronavirus disease pandemic.

This study was designed as a pilot randomised controlled trial with single-blind repeated measures. By using convenience sampling, 36 parents of children with ADHD were recruited from the Parent Resource Centre of The Salvation Army (Centre), a Non-government Organization in Hong Kong, between July to August 2022. Centre staff invited parents of children aged 3-12 diagnosed with ADHD who can communicate and understand Cantonese to participate. Parents who had physical or severe intellectual disabilities, mental disorders or received any form of psychological intervention or psychiatric services were excluded from this study. All eligible parents were randomized to either the intervention group (n=18) or the usual care group (control) (n=18).

Parents assigned to the intervention group received the MBSR programme and usual services from the Centre. MBSR had eight weekly sessions of 2.5 hours each, plus a whole day retreat in small groups between session 6 and 7. The usual care group remained with usual support from the Centre, with interest activities such as cooking classes or calligraphy classes, but without any other form of intervention during this period.

ELIGIBILITY:
Inclusion Criteria:

* parents who have a child aged 3-12 with a confirmed diagnosis of ADHD with or without medications
* able to communicate and understand Cantonese

Exclusion Criteria:

* having physical disabilities or severe intellectual impairments
* any forms of mental disorders
* receiving any other form of psychological intervention, behavioural treatment, or psychiatric services

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Self-report of parental stress | immediate after intervention
  self-report of parental stress as measured by Parental Stress Scale (score range from 1-90. The higher the score, the higher the stress level)
self-report perceived stress | immediate after intervention
  self-report perceived stress as measured by Perceived Stress Scale (score range from 0-56. The higher the score, the higher the stress level)

SECONDARY OUTCOMES:
self-report mindfulness in parenting | At one month after intervention
  Parental self-reports of adopting mindful parenting strategies as measured by Interpersonal mindfulness in Parenting (Score range from 1-155. The higher score means adopted more mindful in parenting)
Parent reports of children's ADHD behaviors in the past 6 months | At one month after intervention
  parent reports of children's ADHD symptoms by using the Strengths and Weakness of ADHD symptoms and normal behavior rating scales (score range from +3 far below average to -3 far above average)
self-report quality of life | At one month after intervention
  self-report to access perception of quality of life in four domains including physical, psychological, social relationships and general health (score range from 0 - 100. A higher score indicated a better quality of life)

CONTACTS AND LOCATIONS:
Overall Officials: Yim Wah MAK, Ph.D, Principal Investigator — School of Nursing, The Hong Kong Polytechnic University
Locations (1):
- The Salvation Army - Hong Kong and Macau Command, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Law TY, Bressington D, Ruan J, Wong WK, Mak YW. The effectiveness of a mindfulness-based stress reduction (MBSR) programme for parents of children with attention deficit hyperactivity disorder (ADHD): a pilot randomized controlled trial. BMC Psychol. 2025 Apr 24;13(1):429. doi: 10.1186/s40359-025-02747-4. PMID 40275428